CLINICAL TRIAL: NCT02985203
Title: A Clinical Study to Investigate the Efficacy and Safety of Combination of Oral Navelbine and Cisplatin Followed by Metronomic Oral Navelbine in Patients With Advanced Non-Small Cell Lung Cancer
Brief Title: Oral Navelbine and Cisplatin Followed by Metronomic Oral Navelbine in Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: No participants were enrolled as schedule.
Sponsor: Guangdong Association of Clinical Trials (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTONG 1512
Record Dates: First submitted 2016-11-29; First posted 2016-12-07 (Estimated); Last update posted 2020-03-12 (Actual); Status verified 2018-06

CONDITIONS: Lung Neoplasm Malignant
Keywords: lung cancer; vinorelbine; metronomic chemotherapy
MeSH Terms: conditions — Lung Neoplasms | interventions — Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vinorelbine oral (Experimental): Oral Navelbine plus Cisplatin followed by metronomic oral vinorelbine.
  Interventions: Drug: Vinorelbine Oral
- Physician's choice (No Intervention): Observation or maintenance therapy other than orla navelbine.

INTERVENTIONS:
Drug: Vinorelbine Oral — Oral vinorelbine plus cisplatin Followed by Metronomic oral Vinorelbine
  Other Names: Navelbine
  Arms: Vinorelbine oral

SUMMARY:
This is an open-label, multi-center clinical trial, aims to evaluate the efficacy and safety of combination of oral Navelbine and Cisplatin followed by metronomic oral Navelbine in Patients with advanced Non-Small Cell Lung Cancer.

The study comprises two stages. In the 1st stage (Week 1-12), all patients will receive combination chemotherapy. In the 2nd stage (Week 13-25), patients who complete the combination chemotherapy with acceptable tolerance and have no progressive disease (PD) will be allocated into 2 arms, to evaluate the efficacy and safety of maintenance chemotherapy with metronomic oral Navelbine (Arm A) or other regimen (Arm B).

DETAILED DESCRIPTION:
In the 1st stage (Week 1-12), all patients will receive combination chemotherapy, i.e. Platinum and Navelbine, for 4 cycles. The regimen is:

Navelbine oral 60mg/m2 d1,8 the first cycle; oral 80mg/m2 day1,8 in sequential cycles q3w plus cisplatin: 75mg/m2 d1 q3w.

In the 2nd stage (Week 13-25), patients who complete the combination chemotherapy with acceptable tolerance and have no PD will be allocated into 2 arms, to evaluate the efficacy and safety of maintenance chemotherapy with metronomic oral Navelbine (Arm A) or other regimen (Arm B). The allocation will be done in sequence at each site, i.e., the first subject who complete the combination chemotherapy with acceptable tolerance and have no PD will be allocated to Arm A, and the second will be allocated to Arm B, and so on. Arm A will continue with oral Navelbine 3 times weekly as maintenance therapy, up to 12 weeks, or till progression, unacceptable toxicity or death occurred. As contrast, Arm B will receive other therapy as per the physician's choice.

Arm A: Navelbine oral 50mg three times per week (Day 1, 3, 5 of each week ) Arm B: Physician's choice (other than Navelbine oral) computed tomography (CT) or magnetic resonance imaging (MRI) will be done at the screening visit, Week 7, Week 13 (before the initiation of maintenance therapy), Week 19 (after 6 weeks of maintenance therapy), and Week 25 (after 12 weeks of maintenance therapy), to evaluate the tumor response. The Disease Control Rate (proportion of patients in complete response (CR), partial response (PR) or stable disease (SD)) after 6 weeks and 12 weeks of maintenance therapy will be evaluated separately for the 2 arms. And Arm B is for observational study only, and will provide rationale for control group selecting in future study.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged ≥ 18 years with life expectancy ≥ 6 months
* Histologically or cytologically confirmed advanced (Stage III B - IV) NSCLC which has not received antineoplastic treatment and not suitable for radical treatment, including those have been resected more than 1 year before signing informed consent form (ICF) then metastasized or relapsed and currently requiring chemotherapy
* With no history of cancer other than in situ uterine cervix cancer or skin basal cell carcinoma with no active disease within 5 years prior to signing the ICF
* With at least one measurable target lesion(s) according to RECIST 1.1
* Adequate hematopoietic function
* Adequate hepatic and renal function
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-1
* Women of child-bearing potential must have a negative pregnancy test (urine or serum) within 7 days of drug administration and agree to take an adequate contraceptive measure
* Men who have sexual life and have a wife of child-bearing age must agree to take an adequate contraceptive measure during and for 12 weeks after the last treatment with Navelbine
* Signed written informed consent
* Able to comply with the protocol

Exclusion Criteria:

* Non-small Cell Lung Cancer with positive sensitizing epidermal growth factor receptor (EGFR) mutation positive or anaplastic lymphoma kinase (ALK) fusion oncogene, or with unknown EGFR/ALK status
* Resectable Non-Small Cell Lung Cancer or suitable for radical radiotherapy/ chemotherapy
* Patients with medical conditions that the only manifestation is hydrothorax, ascites, bone lesions or other unmeasurable diseases
* Symptomatic CNS metastasis (CNS metastasis which has received radiotherapy or surgery and symptom has been stable for more than 4 weeks could be enrolled)
* With invasive malignancies except lung cancer
* Inadequate hematopoietic function:

  * Neutrophil <1.5*109/L;
  * Hb < 100g/L;
  * platelet count (PLT) <100*109/L
* Inadequate hepatic or renal function:

  * aspartate aminotransferase (AST)/alanine aminotransferase (ALT)/alkaline phosphatase (AKP)>2.5 upper limit of normal (ULN) in patients without liver or bone metastasis
  * AST and/or ALT >1.5 ULN with AKP>2.5 ULN
  * AKP>5 ULN in patients with bone metastasis
  * ALT/AST>5 ULN in patients with liver metastasis
  * Total bilirubin > 1.5 ULN
  * Serum creatinine >1.5 ULN
  * Calculated creatinine clearance below 60ml/min (Cockcroft and Gault formula)
  * Blood calcium>ULN
* Patient is pregnant or nursing
* Patients with psychiatric disorder or other disease leading to incompliance to the therapy
* Known hypersensitivity to any ingredient of the regimen
* Treatment with any investigational drug within 30 days before the beginning of treatment with study drug
* Malabsorption syndrome or any other disorder affecting gastrointestinal absorption
* Any other severe, acute, or chronic medical condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration or may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the patient inappropriate for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2016-11; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Disease control rate during maintenance | 12 weeks

SECONDARY OUTCOMES:
Response rate during maintenance | 12 weeks
Duration of response | 8 months
progression-free survival | 8 months

OTHER OUTCOMES:
Adverse events | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Zhen Wang, PhD,MD, Principal Investigator — Guangdong General Hospital&Guangdong Academy of Medical Sciences
Locations (1):
- Guangdong General Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No